CLINICAL TRIAL: NCT02691858
Title: Effect of Hydrocortisone on Improving Outcome of Pneumatic Reduction of Infantile Intussusception: A Randomized Controlled Trial
Brief Title: Effect of Hydrocortisone on Improving Outcome of Pneumatic Reduction of Infantile Intussusception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud El Fiky, Lecturer of Pediatric Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIUNIPEDSURG-CR3
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Intussusception
Keywords: Intussusception
MeSH Terms: conditions — Intussusception | interventions — Hydrocortisone; hydrocortisone hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrocortisone (Experimental): Hydrocortisone IV 10 mg/kg with Resuscitation before attempting reduction, single dose with Resuscitation before attempting reduction
  Interventions: Drug: Hydrocortisone
- Saline (Placebo Comparator): Saline IV 100 ml with Resuscitation before attempting reduction, single dose with Resuscitation before attempting reduction
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Hydrocortisone — 10 mg/kg with Resuscitation before attempting pneumatic reduction, single dose with Resuscitation before attempting reduction
  Other Names: Solu-Cortef
  Arms: Hydrocortisone
Drug: Saline — 100 ml with Resuscitation before attempting pneumatic reduction, single dose with Resuscitation before attempting reduction
  Other Names: sodium chloride 0.9%
  Arms: Saline

SUMMARY:
Intussusception is one of the most frequent causes of acute bowel and second most common cause of acute abdominal pain in pediatric age .95 % of cases are idiopathic, the rest are either due to pathological lead point or post operative. Treatment of intussusception must start with medical resuscitation, then radiological or operative reduction of intussusception.

Our surgery team has used hydrocortisone with the medical resuscitation to improve the success rate of pneumatic reduction and decrease the number of reduction trials.

DETAILED DESCRIPTION:
Experimental group will be given single dose IV Hydrocortisone 10 mg/kg with Resuscitation before attempting first trial of pneumatic reduction and the outcome measured.

Control group will be given Saline 100 ml IV single injection with Resuscitation before attempting first trial of pneumatic reduction and the outcome measured.

ELIGIBILITY:
Inclusion Criteria:

* Infantile Intussusception

Exclusion Criteria:

* Peritonitis Pneumoperitoneum Morbid patients

Ages: 3 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Success of Pneumatic Reduction | 1 Hour
  Comparing number of Successful Pneumatic Reductions in both groups

SECONDARY OUTCOMES:
Reducing number of trials of Pneumatic Reduction | 2 Hours
  Comparing average number of Pneumatic Reduction trials between both groups
Reducing complications | 2 Hours
  Comparing number of complications in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Gamal El Tagy, MD, Study Chair — Cairo University
Locations (1):
- Cairo University Pediatric Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gersema, Lisa, and Karen Baker.
- [Result] Kara, Cüneyt Orhan, and Inci Gökalan.